CLINICAL TRIAL: NCT01824264
Title: A Multi-center, Randomized, Double-blind, Parallel-group Dose-finding Study to Evaluate Change in HbA1c After 12 Weeks Monotherapy With 7 Doses of LIK066 Compared With Placebo or Sitagliptin in Patients With Type 2 Diabetes
Brief Title: Dose-finding Study of LIK066 Compared With Placebo or Sitagliptin to Evaluate Change in HbA1c in Patients With Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIK066A2202; 2012-005793-63 (EudraCT Number)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes mellitus, SGLT inhibitors, dose-response
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — licogliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- LIK066 2.5 mg (Experimental): Patients receive 2.5 mg of LIK066 once daily for 12 weeks
  Interventions: Drug: LIK066
- LIK066 5 mg (Experimental): Patients receive 5 mg of LIK066 once daily for 12 weeks
  Interventions: Drug: LIK066
- LIK066 10 mg (Experimental): Patients receive 10 mg of LIK066 once daily for 12 weeks
  Interventions: Drug: LIK066
- LIK066 25 mg (Experimental): Patients receive 25 mg of LIK066 once daily for 12 weeks
  Interventions: Drug: LIK066
- LIK066 50 mg (Experimental): Patients receive 50 mg of LIK066 once daily for 12 weeks
  Interventions: Drug: LIK066
- LIK066 100 mg (Experimental): Patients receive 100 mg of LIK066 once daily for 12 weeks
  Interventions: Drug: LIK066
- LIK066 150 mg (Experimental): Patients receive 150 mg of LIK066 once daily for 12 weeks
  Interventions: Drug: LIK066
- Sitagliptin 100 mg (Active Comparator): Patients receive 100 mg sitagliptin once daily for 12 weeks
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Patients receive placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIK066 — Experimental treatment doses
  Arms: LIK066 10 mg; LIK066 100 mg; LIK066 150 mg; LIK066 2.5 mg; LIK066 25 mg; LIK066 5 mg; LIK066 50 mg
Drug: Sitagliptin — Active comparator treatment dose
  Arms: Sitagliptin 100 mg
Drug: Placebo — Placebo comparator dose
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy, tolerability and short-term safety of LIK066 to support dose selection for phase 3.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of T2DM by standard criteria
2. Drug-naïve patients, defined as patients not having received any anti-diabetic medication previously,
3. Currently untreated patients , who, after the diagnosis of T2DM, have received anti-diabetic medication for not more than 12 consecutive weeks, and have not received any anti-diabetic treatment within 12 weeks prior to Visit 1
4. Patients being treated with mono-therapy for at least 8 consecutive weeks prior to Visit 1 with the following OADs: metformin, dipeptidyl peptidase-4 inhibitors (DPP-4i), SU, glinide, alpha-glucosidase inhibitor (AGI)
5. HbA1c ≥ 7 to ≤ 10.5% at Visit 1 for drug-naïve/currently untreated patients
6. HbA1c ≥ 7 to ≤ 9.5% at Visit 1 for patients treated with OAD monotherapy
7. HbA1c ≥ 7 to ≤ 10.5% at Visit 199 for ALL patients
8. Age: ≥18 and ≤ 75 years old at Visit 1
9. BMI ≥22 to ≤45 kg/m2 at Visit 1

Exclusion Criteria:

1. FPG ≥270 mg/dl (15 mmol/L) for drug-naïve/currently untreated patients or ≥240 mg/dl (13.3 mmol/L) for patients on OAD monotherapy at Visit 1
2. Insulin treatment >4 consecutive weeks in the last 6 months, corticosteroid use >7 days in the last 8 weeks, use of growth hormones in the last 6 months, or use of weight control products > 4 weeks in the last 6 months
3. History of acute metabolic complications, CV disease, type 1 diabetes mellitus, hepatic disorders, pancreatitis, chronic diarrhea
4. Significant lab abnormalities such as TSH outside of normal range, UACR>300 mg/g creatinine, eGFR <60 ml/min/1.73m2, hemoglobin <12 g/L in men and <11 g/L in women, hematuria
5. ECG abnormalities including AV block, long QT syndrome or QTc>450 msec for men and >470 msec for women
6. History of malignancy
7. Women of child-bearing potential not using effective methods of contraception Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in glycated hemoglobin (HbA1c) after 12 weeks | baseline, 12 weeks
  Change from baseline in HbA1c after 12 weeks of treatment in each of the LIK066 doses and placebo

SECONDARY OUTCOMES:
Change from baseline in Fasting Plasma Glucose | baseline, 12 weeks
  The effect of LIK066 on fasting plasma glucose after 12 weeks of treatment will be evaluated.
Change from baseline in urinary glucose to creatinine ratio | baseline, 12 weeks
  The effect of LIK066 on urinary glucose to creatinine ratio after 12 weeks of treatment will be evaluated
Change from baseline in Body weight | baseline, 12 weeks
  The effect of LIK066 on change in body weight after 12 weeks of treatment will be evaluated.
Change from baseline in Blood pressure | baseline, 12 weeks
  The effect of LIK066 on change in systolic and diastolic blood pressure after 12 weeks of treatment will be evaluated.
Change from baseline in postprandial glucose during a meal test | baseline, 12 weeks
  The effect of LIK066 on change in postprandial glucose during a meal test after 12 weeks of treatment will be evaluated.
Change from baseline in beta cell function during a meal test | baseline, 12 weeks
  The effect of LIK066 on change in beta cell function during a meal test after 12 weeks of treatment will be evaluated.
Change from baseline in insulin secretion relative to glucose during a meal test | baseline, 12 weeks
  The effect of LIK066on change in insulin secretion relative to glucose during a meal test after 12 weeks of treatment will be evaluated.
Change from baseline in oral glucose insulin sensitivity during a meal test | baseline, 12 weeks
  The effect of LIK066 on change in oral glucose insulin sensitivity during a meal test after 12 weeks of treatment will be evaluated.
Change from baseline in glucagon-like peptide response during a meal test | baseline, 12 weeks
  The effect of LIK066 on change in glucagon-like peptide during a meal test after 12 weeks of treatment will be evaluated.
Change from baseline in Peptide YY response during a meal test | baseline, 12 weeks
  The effect of LIK066 on change in peptide YY response during a meal test after 12 weeks of treatment will be evaluated.
Number of patients with adverse events to assess safety and tolerability of LIK066 | 12 weeks
  The safety and tolerability of 7 doses of LIK066 after 12 weeks of treatment will be evaluated with number of patients reported for total adverse events, serious adverse events and death.
Change from baseline in renal threshold for glucose excretion | baseline, 12 weeks
  The effect of LIK066 on renal threshold for glucose excretion will be calculated from glucose values in an overnight urine collection

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals